CLINICAL TRIAL: NCT07099768
Title: Correlation Between the Flexibility of Hip Muscles, Pain and Disability in Chronic Nonspecific Low Back Pain
Acronym: NSLBP
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shimaa Rabie Tony Mohamed, Principal investigator: Shimaa Rabie Tony Mohamed, Cairo University
Other Study IDs: P.T.REC/012/005813
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Non Specific Low Back Pain
Keywords: Correlation; Flexibility of Hip Muscles; Pain; Disability; Nonspecific Low Back Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 50 subjects aged between 20 and 45 years of both sexes with diagnosis of nonspecific low back pain

SUMMARY:
This study will be conducted to investigate the correlation between the flexibility of hip muscles; hip flexors (iliopsoas, rectus femoris), hip extensors (hamstring), hip internal rotators, hip external rotators, hip adductors and hip abductors with pain intensity and disability level among patients with chronic nonspecific low back pain

DETAILED DESCRIPTION:
Low back pain is considered the primary cause of disability worldwide. Low back pain is pain located at the area from the last ribs to the gluteal region with or without radiation to the lower limbs. Low back pain is associated with substantial economic burden, resulting from healthcare expenses, reduced productivity, insurance costs and sick leaves.

It was reported that limitation of hip range of motion of low-back pain patients was significantly different from that of healthy person. Due to the anatomic proximity and muscle connections, a number of studies have investigated the relationship between hip mobility and episodes of low back pain. From biomechanical point of view limited hip range of motion is compensated by hypermobility of the lumbar region thus generating overload with repetitive compensatory movements in the back.

Patients with non-specific low back pain demonstrate alteration in hip muscles flexibility. This relationship is important because the hip muscles act as an important link between the lower limbs and the trunk exerting forces from the lower limbs to the spine as well as from the spine. Any flexibility limitations of hip muscles not only decreases the range of motion but can also cause excessive mechanical stresses to lumbar spine during particular movement, thus affecting gait and other functional movements.

Up to the author's knowledge, there is few studies that investigates the correlation between the flexibility of all hip muscles and pain intensity and disability level in nonspecific low back pain patients. Therefore, this study aims to assess the correlation between the flexibility of hip muscles; hip flexors (iliopsoas, rectus femoris), hip extensors (hamstring), hip internal rotators, hip external rotators, hip adductors and hip abductors with pain intensity and disability among patients with chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic nonspecific low back pain for at least 3 months.
* Age of the patient will range from 20 and 45 years.
* Pain intensity of three or higher based on the visual analogue scale (VAS, 0-10 scale).
* .Body Mass Index from 18-25 kg/m2.

Exclusion Criteria:

* spinal surgery, spinal or pelvic fracture.
* ankylosing spondylitis or rheumatoid arthritis.
* spondylolisthesis or spondylolysis, neurological disorders.
* spinal inflammation or tumor. osteoporosis.
* Continuous use of pain medications.
* respiratory disease or heart disease.
* Pregnancy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 patients with chronic non specific low back pain from both gender will participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Flexibility of Hip Muscles | up to 1 day
  Flexibility of the muscles of hip will be conducted on both the right and lift side and will be measure by universal Goniometer
Pain Intensity | up to 1 day
  Visual analog scale is globally used as a measure of pain intensity. Visual analogue scale is the most frequent outcome tools in musculoskeletal pain assessment. An overall score between 0 and 10 points is given, with 'no pain' defined as 0 points and 'the most severe pain possible' defined as 10 points.
Disability | up to 1 day
  Oswestry disability index is an internally consistent, unidimensional scale with overall excellent construct validity and ability to discriminate the severity of functional disability. The analysis suggests that the Oswestry disability index may better distinguish between the relative degrees of function at above-average disability levels. The Oswestry disability index is used to assess the extent of disability caused by low back pain, The Oswestry disability index consists of 10 questions on pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual activity, social life, and travel. Performance in each item is described in 6 stages, from 0 to 5 points, A higher score on the Oswestry disability index indicates more severe disability